CLINICAL TRIAL: NCT05354167
Title: Comparison of Muscle Energy Technique and Oscillating Energy Manual Therapy in Chronic Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01053 Huma mehrin
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Lateral Epicondylitis
Keywords: lateral epicondylitis; Muscle energy technique; Oscillating manual energy therapy; grip strength; pain
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- muscle energy technique (Experimental): the subject to sit comfortably and then stabilize the subject's distal humerus with one hand, then the forearm was supinated with the therapist another hand until resistance appeared. Holding the position the subject was asked to slowly pronate the forearm that is Isometric contraction against resistance for a period of 6-10 seconds with inhale and exhale, followed by slightly increasing supination until resistance was met once again. After 5 seconds of relaxation, the procedure was repeated 5 times during a single treatment session.
  Interventions: Other: muscle energy technique
- oscillating manual energy therapy (Experimental): It is also known as V-spread .The subject was asked to sit on a chair with the affected painful arm resting on the treatment table. Tender points were palpated. Then the therapist places the index and middle fingers of one hand in a V-shape around the tender point and placed the index finger of the other hand in the medial side of the elbow, diagonally across the located tender point. Gentle pressure was applied a few times using fingertips to the tissues alternatively from the medial and lateral sides to start the oscillations. On the initiation of oscillations, the application of pressure should be stopped and allow the oscillations to continue between the two points of contact on the subject's elbow. This technique was repeated until there were no tender points on palpation. The duration varied from 30 seconds to 2 minutes.
  Interventions: Other: oscillating manual energy therapy

INTERVENTIONS:
Other: muscle energy technique — the subject to sit comfortably and then stabilize the subject's distal humerus with one hand, then the forearm was supinated with the therapist another hand until resistance appeared. Holding the position the subject was asked to slowly pronate the forearm that is Isometric contraction against resistance for a period of 6-10 seconds with inhale and exhale, followed by slightly increasing supination until resistance was met once again. After 5 seconds of relaxation, the procedure was repeated 5 times during a single treatment session; this technique was applied in 2 sessions for a week for 4 weeks.
  Arms: muscle energy technique
Other: oscillating manual energy therapy — It is also known as V-spread .The subject was asked to sit on a chair with the affected painful arm resting on the treatment table. Tender points were palpated. Then the therapist places the index and middle fingers of one hand in a V-shape around the tender point and placed the index finger of the other hand in the medial side of the elbow, diagonally across the located tender point. Gentle pressure was applied a few times using fingertips to the tissues alternatively from the medial and lateral sides to start the oscillations. On the initiation of oscillations, the application of pressure should be stopped and allow the oscillations to continue between the two points of contact on the subject's elbow.
  Arms: oscillating manual energy therapy

SUMMARY:
Lateral epicondylitis (LE) is a painful musculoskeletal condition caused by overuse. The condition is also called tennis elbow because it affects 50% of tennis players, notably beginners learning the one-handed backhand. Nonetheless, only 10% of all patients with LE play tennis. Lateral Epicondylitis (LE) or tennis elbow affects about 1-3% of general population.

Muscle energy technique was developed by osteopathic physician, Fred Mitchell, Sr. It was refined and systematized by Fred Mitchell, Jr., and has continued to evolve with contributions from many individuals.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is a painful musculoskeletal condition caused by overuse. The condition is also called tennis elbow because it affects 50% of tennis players, notably beginners learning the one-handed backhand. Nonetheless, only 10% of all patients with LE play tennis. Lateral Epicondylitis (LE) or tennis elbow affects about 1-3% of general population.

patients with Lateral Epicondylitis complains of pain, functional difficulty affecting activities of daily living related to wrist and forearm movements . The grip strength is affected due to voluntary decline of effort to avoid pain and due to wasting of affecting muscles seen in long standing conditions. The symptoms exacerbate with stressful activities in overuse syndromes but pain may persist even at rest as the condition progress.

Muscle energy technique was developed by osteopathic physician, Fred Mitchell, Sr. It was refined and systematized by Fred Mitchell, Jr., and has continued to evolve with contributions from many individuals. Muscle energy technique (MET) is used by practitioners from different professions and has been advocated for the treatment of shortened muscles, weakened muscles, restricted joints, and lymphatic drainage. In addition to using muscle effort to mobilize joints and tissues, MET is considered by some to be a biomechanics-based analytic diagnostic system that uses precise physical diagnosis evaluation procedures to identify and qualify articular range of motion restriction. MET are defined as a manual treatment in which a patient produces a contraction in a precisely controlled position and direction against a counterforce applied by a manual therapist. MET have been also used in asymptomatic subjects in order to increase mobility. There is varying evidence that when a joint has a functional limitation, the application of a MET can increase its Range of Motion.

A comparative study concluded that oscillating energy manual therapy and muscle energy technique had shown the improvement in Numeric Rating Scale, grip strength and PRTEE in lateral epicondylitis subjects, but more significant improvement was observed in the subjects who were treated with muscle energy technique than oscillating energy manual therapy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of tenderness point on lateral epicondyle.
* Positive cozen test, mills test, Maudsley's test
* Negative Radial nerve test

Exclusion Criteria:

* Cervical spine disorder
* Peripheral neuropathy
* Fractures
* Major upper limb surgery
* Steroid injections in last 6 months
* Tumor or wound
* take any kind of physiotherapy treatment

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale | four weeks
  The Verbal Numerical Rating Scale is the most commonly used self-report measure of pain intensity. Patients are instructed to choose a single number from the scale that best indicates their level of pain.1-4 Mild pain,5-6 Moderate,7-10 severe. assessment to be done on baseline and after every week
Hand dynamometer(Grip strength) | for four weeks
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength. Assessment to be done on baseline and after every week.
Patient rated tennis elbow evaluation (functional status) | for four weeks
  The Patient-rated Tennis Elbow Evaluation (PRTEE) enables quantitative rating by the patient of pain and functional impairment associated with tennis elbow or lateral elbow tendinopathy. It takes the form of a 15-item questionnaire, with five items addressing pain and 10 concerned with functional deficit. Assessment to be done on baseline and after every week.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- National Institute of Rehabilitation Medicine,, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No